CLINICAL TRIAL: NCT01383369
Title: Postoperative Sleep Disturbances Role in Cognitive Test Results After Fast-track Hip and Knee Arthroplasty
Status: Completed | Type: Observational
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Lene Krenk, Doctor, Rigshospitalet, Denmark
Other Study IDs: H-C-FSP-2010-050
Record Dates: First submitted 2011-06-23; First posted 2011-06-28 (Estimated); Last update posted 2011-09-28 (Estimated); Status verified 2011-09

CONDITIONS: Postoperative Cognitive Abilities

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The purpose of this study is to evaluate sleep cycle before and after fast-track arthroplasty (3 days before and 10 days after) combined with cognitive testing preoperatively, on postoperative day 1,2,10.

ELIGIBILITY:
Inclusion Criteria:

* above 60
* ASA classification I-IV

Exclusion Criteria:

* general anaesthesia within 90 days
* daily use of sedatives, hypnotics og anxiolytics
* alcohol abuse
* insufficient written and verbal Danish
* severe hearing loss and poor sight
* Parkinsons Disease or other functional neurological deficits
* Mini mental status < 24
* Shift work

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients above 60 years undergoing hip/knee replacement surgery in a fest track set-up.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2011-02; Primary Completion 2011-08 (Actual); Study Completion 2011-08 (Actual)

PRIMARY OUTCOMES:
Stroop colour word test result on the first postoperative morning compared to preoperatively. | 4 days on average between preoperative and postoeperative testing

CONTACTS AND LOCATIONS:
Overall Officials: Lene Krenk, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Gentofte Hospital, Hellerup, Denmark